CLINICAL TRIAL: NCT03657771
Title: A Food Additive Removal Diet for Pediatric Eosinophilic Esophagitis
Acronym: FREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Edward Mougey, Research Scientist, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1173700
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Eosinophilic Esophagitis
Keywords: Esophagitis; Diet
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis

STUDY DESIGN:
Intervention Model Description: Randomized, prospective, parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DED (Active Comparator): Diet eliminating dairy
  Interventions: Other: DED
- FREE (Active Comparator): Diet eliminating dairy and food additives
  Interventions: Other: FREE

INTERVENTIONS:
Other: DED — DED: Diet eliminating dairy
  Arms: DED
Other: FREE — FREE: Diet eliminating dairy and food additives
  Arms: FREE

SUMMARY:
Prospective, pragmatic standard of care clinical trial comparing dietary therapies of standard dairy elimination diet alone (DED) to dairy elimination plus food additive elimination (FREE)

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) is a chronic inflammatory disorder of the esophagus. Primary symptoms manifest while eating and include dysphagia, chest pain, and food impaction. EoE was first described in the 1990s, but is increasingly recognized worldwide. It affects both adults and children.

Given that EoE is thought to be an allergen driven disease, elimination diets are considered logical and safe first-line treatment options. Elimination diets focus on the removal of the food groups most likely to evoke the inflammatory response (e.g. dairy, wheat, soy, egg, etc.). This is the first study to examine the effects of an additive free diet on eosinophilic esophagitis.

Primary Objective: To compare histologic outcomes (eosinophils per high power field: eos/hpf) of DED and FREE in children with eosinophilic esophagitis.

Secondary Objective: To compare endoscopic outcomes (Eosinophilic Esophagitis Endoscopic Reference scores: EREFs) of DED and FREE in children with eosinophilic esophagitis

Tertiary Objectives: To compare symptomatic (Pediatric Eosinophilic Esophagitis Symptom Severity Module v2.0: PEESS) and quality of life (Peds-QL EoE Module 1) outcomes of DED and FREE in children with eosinophilic esophagitis

The investigators plan to enroll 72 patients over 4 sites each enrolling 18 patients per site in a 16-month period (approximately 1 patient per month per site) having 9 patients per site in each group (DED and FREE).

The investigators will enroll patients > 5- <17 years of age with isolated esophageal eosinophilia (>15 eos/hpf). Patients with food impaction, peripheral eosinophilia > 1,500 µL , concomitant GI inflammatory conditions, history of upper GI tract surgery (e.g. fundoplication), acid reflux by pH probe, anaphylactic food allergies, severe developmental delay, taking recently prescribed inhaled corticosteroids or oral corticosteroids, have other medical conditions likely interfere with the study, has a significant psychiatric condition, has taken a PPI in the last 4 weeks, has taken swallowed steroids in the last 12 weeks, or are not fluent in spoken and written English will be excluded.

Participants will be enrolled at: Nemours Children's Hospital, Orlando, FL; Alfred I Dupont Hospital, Wilmington, DE; Seattle Children's Hospital, Seattle, WA

Once eligibility criteria are met, participants will be randomized to DED or FREE study groups. Participants will receive dietary education. Lead dietitians from each site will be identified and the approaches to dietary education will be standardized. Dietary education will be completed at the baseline visit and during follow up phone calls throughout the study.Each participant will complete all study visits in 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB) approved written Parental Permission form is signed and dated by the parent or legal representative/caregiver.
2. If applicable, an Institutional Review Board (IRB) approved written Assent form is signed and dated by the participant.
3. The participant/parent(s) or legal representative(s)/caregiver(s) are considered reliable and capable of adhering to the protocol call schedule and dietary requirements.
4. The participant is >2 years to <18 years of age.
5. The participant has isolated esophageal eosinophilia (>15 eos/hpf).
6. The family has access to the internet to complete weekly surveys and to a telephone to complete weekly follow up calls.
7. The biopsy used to diagnose eosinophilic esophagitis was taken no more than 12 weeks prior to the date of enrollment.

Exclusion Criteria:

1. The participant has peripheral eosinophilia > 1,500 µL
2. The participant has concomitant GI inflammatory conditions (e.g. celiac disease, inflammatory bowel disease).
3. The participant has a history of upper GI tract surgery (e.g. fundoplication)
4. Acid reflux by pH probe is suggested (*A pH probe is not required, but may be done as standard of care)
5. The participant has severe developmental delay that, in the opinion of the investigator, could jeopardize the participant's ability to participate in the study.
6. The participant has taken prednisone in the last 12 weeks, or has taken fluticasone or budesonide in the last 8 weeks.
7. The participant has other significant medical conditions that, in the opinion of the provider, would impact the participant's ability to participate in the study.
8. The participant has a psychiatric condition that, in the opinion of the investigator, could jeopardize the participant's ability to participate in the study.
9. The participant does not speak or read English fluently.
10. The participant is currently taking a PPI (If discontinued, no washout required.)
11. The participant is currently on or previously failed a dairy free diet for EoE.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Eosinophils Per High Power Field (eos/hpf) | 12 weeks
  Histologic change differences of maximum eosinophils per high power field

SECONDARY OUTCOMES:
Eosinophilic Esophagitis Endoscopic Reference Score (EREFS) | 12 weeks
  An endoscopic outcome measure to follow response to treatment. Scores range from 0 to 15 with higher scores indicating more endoscopic evidence of eosinophilic esophagitis.

OTHER OUTCOMES:
Pediatric Eosinophilic Esophagitis Symptom Severity Module (PEESS) | Baseline, 4, 8, and 12 weeks
  Self report measure of symptoms associated with eosinophilic esophagitis. Scores range from 0 to 100. The higher the score, the more frequent and severe the symptoms.
Pediatric Eosinophilic Esophagitis Symptom Severity Module (PEESS): Parent Report | Baseline, 4, 8, and 12 weeks
  Parent report measure of symptoms associated with eosinophilic esophagitis. Scores range from 0 to 100. The higher the score, the more frequent and severe the symptoms.
Pediatric Quality of Life Inventory: Eosinophilic Esophagitis Module (PedsQL-EoE) | Baseline, 4, 8, and 12 weeks
  Self report measure of quality of life and symptoms associated with eosinophilic esophagitis. This measure has several subscales (Symptoms I, Symptoms II, Treatment, Worry, Communication, Food and Eating, Food Feelings) that produce scaled scores ranging from 0 to 100. The total scaled score also ranges from 0 to 100. A higher score indicates better quality of life.
Pediatric Quality of Life Inventory: Eosinophilic Esophagitis Module (PedsQL-EoE): Parent Report | Baseline, 4, 8, and 12 weeks
  Parent report measure of quality of life and symptoms associated with eosinophilic esophagitis. This measure has several subscales (Symptoms I, Symptoms II, Treatment, Worry, Communication, Food and Eating, Food Feelings) that produce scaled scores ranging from 0 to 100. The total scaled score also ranges from 0 to 100. A higher score indicates better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Edward B. Mougey, PhD, Principal Investigator — Nemours Children's Clinic
Locations (3):
- United States (3):
  - Nemours/Alfred I DuPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Hospital, Orlando, Florida
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franciosi JP, Hommel KA, Bendo CB, King EC, Collins MH, Eby MD, Marsolo K, Abonia JP, von Tiehl KF, Putnam PE, Greenler AJ, Greenberg AB, Bryson RA, Davis CM, Olive AP, Gupta SK, Erwin EA, Klinnert MD, Spergel JM, Denham JM, Furuta GT, Rothenberg ME, Varni JW. PedsQL eosinophilic esophagitis module: feasibility, reliability, and validity. J Pediatr Gastroenterol Nutr. 2013 Jul;57(1):57-66. doi: 10.1097/MPG.0b013e31828f1fd2. PMID 23478422
- [Background] Martino JV, Van Limbergen J, Cahill LE. The Role of Carrageenan and Carboxymethylcellulose in the Development of Intestinal Inflammation. Front Pediatr. 2017 May 1;5:96. doi: 10.3389/fped.2017.00096. eCollection 2017. PMID 28507982
- [Background] Dellon ES, Jensen ET, Martin CF, Shaheen NJ, Kappelman MD. Prevalence of eosinophilic esophagitis in the United States. Clin Gastroenterol Hepatol. 2014 Apr;12(4):589-96.e1. doi: 10.1016/j.cgh.2013.09.008. Epub 2013 Sep 11. PMID 24035773
- [Background] Dellon ES, Gonsalves N, Hirano I, Furuta GT, Liacouras CA, Katzka DA; American College of Gastroenterology. ACG clinical guideline: Evidenced based approach to the diagnosis and management of esophageal eosinophilia and eosinophilic esophagitis (EoE). Am J Gastroenterol. 2013 May;108(5):679-92; quiz 693. doi: 10.1038/ajg.2013.71. Epub 2013 Apr 9. PMID 23567357
- [Background] Imam T, Gupta SK. Topical glucocorticoid vs. diet therapy in eosinophilic esophagitis: the need for better treatment options. Expert Rev Clin Immunol. 2016 Aug;12(8):797-9. doi: 10.1080/1744666X.2016.1191947. Epub 2016 Jun 13. No abstract available. PMID 27206496
- [Background] Kagalwalla AF, Wechsler JB, Amsden K, Schwartz S, Makhija M, Olive A, Davis CM, Manuel-Rubio M, Marcus S, Shaykin R, Sulkowski M, Johnson K, Ross JN, Riffle ME, Groetch M, Melin-Aldana H, Schady D, Palac H, Kim KA, Wershil BK, Collins MH, Chehade M. Efficacy of a 4-Food Elimination Diet for Children With Eosinophilic Esophagitis. Clin Gastroenterol Hepatol. 2017 Nov;15(11):1698-1707.e7. doi: 10.1016/j.cgh.2017.05.048. Epub 2017 Jun 8. PMID 28603055
- [Background] Newberry C, Lynch K. Can We Use Diet to Effectively Treat Esophageal Disease? A Review of the Current Literature. Curr Gastroenterol Rep. 2017 Aug;19(8):38. doi: 10.1007/s11894-017-0578-5. PMID 28730507
- [Background] Groetch M, Venter C, Skypala I, Vlieg-Boerstra B, Grimshaw K, Durban R, Cassin A, Henry M, Kliewer K, Kabbash L, Atkins D, Nowak-Wegrzyn A, Holbreich M, Chehade M; Eosinophilic Gastrointestinal Disorders Committee of the American Academy of Allergy, Asthma and Immunology. Dietary Therapy and Nutrition Management of Eosinophilic Esophagitis: A Work Group Report of the American Academy of Allergy, Asthma, and Immunology. J Allergy Clin Immunol Pract. 2017 Mar-Apr;5(2):312-324.e29. doi: 10.1016/j.jaip.2016.12.026. PMID 28283156
- [Background] Kagalwalla AF, Sentongo TA, Ritz S, Hess T, Nelson SP, Emerick KM, Melin-Aldana H, Li BU. Effect of six-food elimination diet on clinical and histologic outcomes in eosinophilic esophagitis. Clin Gastroenterol Hepatol. 2006 Sep;4(9):1097-102. doi: 10.1016/j.cgh.2006.05.026. Epub 2006 Jul 21. PMID 16860614
- [Background] Gonsalves N, Yang GY, Doerfler B, Ritz S, Ditto AM, Hirano I. Elimination diet effectively treats eosinophilic esophagitis in adults; food reintroduction identifies causative factors. Gastroenterology. 2012 Jun;142(7):1451-9.e1; quiz e14-5. doi: 10.1053/j.gastro.2012.03.001. Epub 2012 Mar 3. PMID 22391333
- [Background] Suskind DL, Wahbeh G, Gregory N, Vendettuoli H, Christie D. Nutritional therapy in pediatric Crohn disease: the specific carbohydrate diet. J Pediatr Gastroenterol Nutr. 2014 Jan;58(1):87-91. doi: 10.1097/MPG.0000000000000103. PMID 24048168
- [Background] Collins MH, Martin LJ, Alexander ES, Boyd JT, Sheridan R, He H, Pentiuk S, Putnam PE, Abonia JP, Mukkada VA, Franciosi JP, Rothenberg ME. Newly developed and validated eosinophilic esophagitis histology scoring system and evidence that it outperforms peak eosinophil count for disease diagnosis and monitoring. Dis Esophagus. 2017 Feb 1;30(3):1-8. doi: 10.1111/dote.12470. PMID 26857345

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/71/NCT03657771/Prot_SAP_004.pdf
  • Informed Consent Form (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03657771/ICF_005.pdf